CLINICAL TRIAL: NCT02960984
Title: Effects of Neurorehabilitation on Upper Limb Performance and on Fatigue in People With Multiple Sclerosis
Brief Title: Neurorehabilitation on Upper Limb and on Fatigue in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Genova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UL_SM
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurorehabilitation (Experimental): Participants in the experimental group will receive 1 hour treatment comprising 30' of aerobic training on an ergometer and 30' of task-oriented training focused on uppper limb rehabilitation.
  Interventions: Other: Task Oriented rehabilitation and aerobic training
- Baseline (No Intervention): No intervention is planned

INTERVENTIONS:
Other: Task Oriented rehabilitation and aerobic training — Participants in the experimental group will receive 1 hour treatment comprising 30' of aerobic training and 30' of task-oriented training focused on uppper limb rehabilitation for 3 times a week for 20 sessions.
  Arms: Neurorehabilitation

SUMMARY:
In Multiple Sclerosis the multiplicity of physical and psychological dysfunctions have been shown to exhibit a number of life-altering problems such as fatigue, limb weakness, alteration of upper extremity fine motor coordination, loss of sensation, spasticity. These problems affect performance of many daily living activities (ADL) such as dressing, bathing, self-care, and writing, thus reducing functional independence and self-rated quality of life.

Twenty people with Multiple Sclerosis will receive neurorehabilitation treatment comprising a combination of aerobic training and upper limb task-oriented training.

The aim of this pilot crossover study is to evaluate the effects of neurorehabilitation on upper limb performance and on fatigue in People with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* no relapses in the last three months
* Expanded Disability Status Scale (EDSS) ≤ 8;

Exclusion Criteria:

* subjects with relapses
* worsening of the pathology in the last three months
* subjects with cognitive and psychiatric disturbances
* subjects with cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 9-hole peg test at 2 and 4 months | baseline, then participants were followed for the duration the outpatient treatment protocol, an average of 8 weeks, and at follow up 2 months after the end of the treatment protocol
Change from Baseline in Heart Rate at 2 and 4 months | baseline, then participants were followed for the duration the outpatient treatment protocol, an average of 8 weeks, and at follow up 2 months after the end of the treatment protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Gnocchi ONLUS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided